CLINICAL TRIAL: NCT05187663
Title: The Evaluation of Clinical, Microbiological and Immunological Parameters After Using Photodynamic Therapy in the Surgical Treatment of Peri-implantitis: Randomized Clinical Trials.
Brief Title: Evaluation of Photodynamic Therapy in Treatment of Peri-implantitis
Acronym: PDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Collaborators: Military Medical Academy, Bulgaria (Other); Bredent Medical, Helbo (Other)
Responsible Party: Principal Investigator, Dragana Rakasevic, PhD, Specialist of periodontology, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 39/28
Record Dates: First submitted 2021-12-12; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Peri-Implantitis
Keywords: Peri-Implantitis, Photodynamic therapy, Surgery
MeSH Terms: conditions — Peri-Implantitis | interventions — 1-phenyl-3,3-dimethyltriazene; Population Groups; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double (Participant, Investigator, Sub-investigator) Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): In the test group, implant surface decontamination was performed with photodynamic therapy.
  Interventions: Procedure: Photodynamic (PDT) group
- Control group (Active Comparator): In the control group, implant surface decontamination was performed with 1% chlorhexidine gel.
  Interventions: Procedure: Chlorhexidine (CHX) group

INTERVENTIONS:
Procedure: Photodynamic (PDT) group — Mucoperiostal buccal and lingual incisions were made using a surgical blade under local anaesthesia. Full-thickness mucoperiosteal flaps were elevated buccally and lingually. In the photodynamic (PDT) group, after careful removal of granulation tissue and mechanical debridement of the implant surface, decontamination of implant surfaces and peri-implant tissues was performed using the photodynamic therapy, PDT (HELBO, Photodynamic Systems GmbH, Wels, Austria). The implant surface and the surrounding tissue were exposed to the laser light by means of fibres (HELBO ® TheraLite Laser HELBO ® 2D Spot Probe; bredent medical GmbH & Co KG) for the 30s/spot, which operates on the wavelength of 660 nm and irradiance of 100 Mw. Bone augmentation and bio-resorbable membrane were applied in peri-implant defects using the bovine bone substitute and collagen membrane (Bio -Oss and Bio Guide, GeistlichPharma; Dembone). The mucoperiosteal flaps were repositioned and sutured.
  Arms: Study group
Procedure: Chlorhexidine (CHX) group — Mucoperiostal buccal and lingual incisions were made using a surgical blade under local anaesthesia. Full-thickness mucoperiosteal flaps were elevated buccally and lingually. In the chlorhexidine (CHX) group, after careful removal of granulation tissue and mechanical debridement of the implant surface 1% gel of chlorhexidine (Chlorhexamed® - Direkt) was applied on the implant surface for one minute and irrigated for 1 min by saline. Bone augmentation and bio-resorbable membrane were applied in peri-implant defects using the bovine bone substitute and collagen membrane (Bio -Oss and Bio Guide, GeistlichPharma; Dembone). The mucoperiosteal flaps were repositioned and sutured.
  Arms: Control group

SUMMARY:
Photodynamic therapy (PDT) is suggested as an adjuvant treatment method to the surgery in peri-implantitis treatment. The primary goal of peri-implantitis therapy is the removal of the causative bacteria from the implant surface and surrounding tissues in order to improve the process of re-osseointegration and achieve long term implant stability. Accordingly, the aims of the study were to evaluate clinical, immunological and microbiological outcomes after surgical therapy of peri-implantitis following PDT.

DETAILED DESCRIPTION:
Treatment procedure

After clinical parameters were recorded and samples were taken, all patients underwent a single episode of non-surgical therapy. It implied a mechanical method for debridement of implants and remaining dentition in order to reduce signs of inflammation. Instructions for oral hygiene were proposed in the same visit.

Peri-implantitis surgical treatment was conducted by one experienced surgeon two weeks after non-surgical therapy. After granulation tissue removal and mechanical implant surface cleaning with graphite curettes (Straumann Dental Implant System Straumann AG, Basel, Switzerland), decontamination of implant surface was conducted. In the study group, for the decontamination of implant surfaces and peri-implant tissues photodynamic therapy was performed (HELBO, Photodynamic Systems GmbH, Wels, Austria), while in the control group, after removal of granulation tissue, 1% gel of chlorhexidine (Chlorhexamed® - Direkt) was put on the implant surface. One minute after exposing the implant surface with CHX, it was irrigated for 1 min by saline. Bone augmentation and bio-resorbable membrane were applied in peri-implant defects using the bovine bone substitute and collagen membrane (Bio-Oss and Bio Gide, GeistlichPharma; Dembone). The mucoperiosteal flaps were repositioned and sutured [17, 19].

Patients were prescribed antibiotics (Amoxicillin, 500 mg, three per day, 5 days). It was recommended that patients don't use mouthwash during the postoperative period.

Clinical, immunological and microbiological parameters were measured and assessed baseline, three, six, 12 and 24 months postoperatively. Immunological parameters (IL-17, IL-1β, IL-6) were analysed by ELISA while microbiological samples were collected before the therapy, during the surgery, and at follow-up periods.

Assessment of implant macro- and micro- design were additionally assessed.

ELIGIBILITY:
Inclusion Criteria:

1. More than 18 years old
2. No periodontal or peri-implant treatment in the last 3 months prior to the study
3. Presence of a minimum of one implant in function more than one year with signs of early and moderate peri-implantitis
4. Prosthetic rehabilitation of the implant with diagnosed peri-implantitis more than 6 months
5. Presence of peri-implant pocket depth more than 4 mm
6. Radiogrpih bone level loss more than 2 mm 7 Positive sign of bleeding on probing with or without suppuration

Exclusion Criteria:

1. Uncontrolled medical conditions
2. Use of systemic antibiotics in the previous 3 months
3. Use of anti-inflammatory drugs in the previous 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — > 18 years of age
Enrollment: 50 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change of bleeding on probing (BOP) | Change baseline BOP at 12 months
  Evaluated as present if bleeding was evident within 30 s after probing, or absent, if no bleeding was observed
Change of bleeding on probing (BOP) | Change baseline BOP at 24 months
  Evaluated as present if bleeding was evident within 30 s after probing, or absent, if no bleeding was observed

SECONDARY OUTCOMES:
Change of peri-implant probing depths (PPD) | Change baseline PPD at 12 months
  PPD was measured in millimetres as the distance from mucosal margin to bottom of periodontal pocket.
Change of peri-implant probing depths (PPD) | Change baseline PPD at 24 months
  PPD was measured in millimetres as the distance from mucosal margin to bottom of periodontal pocket.
Change of clinical attachment gain (CAG) | Change baseline CAL at 12 months
  CAL, measured in millimetres as the distance from implant shoulder to the bottom of peri-implant pocket at six points.
Change of clinical attachment gain (CAG) | Change baseline CAL at 24 months
  CAL, measured in millimetres as the distance from implant shoulder to the bottom of peri-implant pocket at six points.

OTHER OUTCOMES:
Concentration of interleukin 17 (IL-17) | Change baseline concentration of IL-17 at 12 months
  Measurement of pro-inflammatory IL-17 concentration before and after the treatment procedure.
Concentration of interleukin 17 (IL-17) | Change baseline concentration of IL-17 at 24 months
  Measurement of pro-inflammatory IL-17 concentration before and after the treatment procedure.
Concentration of interleukin 1 beta (IL-1beta) | Change baseline concentration of IL-1beta at 12 months
  Measurement of pro-inflammatory IL-1beta concentration before and after the treatment procedure.
Concentration of interleukin 1 beta (IL-1beta) | Change baseline concentration of IL-1beta at 24 months
  Measurement of pro-inflammatory IL-1beta concentration before and after the treatment procedure.
Concentration of interleukin 6 (IL-6) | Change baseline concentration of IL-6 at 12 months
  Measurement of pro-inflammatory IL-6 concentration before and after the treatment procedure.
Concentration of interleukin 6 (IL-6) | Change baseline concentration of IL-6 at 24 months
  Measurement of pro-inflammatory IL-6 concentration before and after the treatment procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontal and Oral Mucosa Diseases, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Gained results are planned to be published in international journal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 2022. to 2032.
Access Criteria: The investigators will be shared analyzed outcomes and surgical procedure protocols

REFERENCES:
- [Background] Heitz-Mayfield LJA, Salvi GE, Mombelli A, Faddy M, Lang NP. Anti-infective surgical therapy of peri-implantitis. A 12-month prospective clinical study. Clin Oral Implants Res. 2012 Feb;23(2):205-210. doi: 10.1111/j.1600-0501.2011.02276.x. Epub 2011 Aug 9. PMID 22092831
- [Background] Marotti J, Tortamano P, Cai S, Ribeiro MS, Franco JE, de Campos TT. Decontamination of dental implant surfaces by means of photodynamic therapy. Lasers Med Sci. 2013 Jan;28(1):303-9. doi: 10.1007/s10103-012-1148-6. Epub 2012 Jul 12. PMID 22790655
- [Background] Dortbudak O, Haas R, Bernhart T, Mailath-Pokorny G. Lethal photosensitization for decontamination of implant surfaces in the treatment of peri-implantitis. Clin Oral Implants Res. 2001 Apr;12(2):104-8. doi: 10.1034/j.1600-0501.2001.012002104.x. PMID 11251658
- [Background] de Waal YC, Raghoebar GM, Meijer HJ, Winkel EG, van Winkelhoff AJ. Implant decontamination with 2% chlorhexidine during surgical peri-implantitis treatment: a randomized, double-blind, controlled trial. Clin Oral Implants Res. 2015 Sep;26(9):1015-23. doi: 10.1111/clr.12419. Epub 2014 May 26. PMID 24861411
- [Background] Froum SJ, Rosen PS. A proposed classification for peri-implantitis. Int J Periodontics Restorative Dent. 2012 Oct;32(5):533-40. PMID 22754901
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/29652462/ — Rakašević D, Lazić Z, Rakonjac B, Soldatović I, Janković S, Magić M, Aleksić Z. Efficiency of photodynamic therapy in the treatment of peri-implantitis - A three-month randomized controlled clinical trial. Srp Arh Celok Lek. 2016 Sep-Oct;144(9-10):478-84. PMID: 29652462.